CLINICAL TRIAL: NCT03335852
Title: Evaluation of Safety and Systemic Pharmacokinetics After Abicipar Pegol (AGN-150998) Intravitreal Injections in Japanese Patients With NEovascular Age-Related Macular Degeneration (PINE Study)
Brief Title: Safety and Pharmacokinetics of Abicipar Pegol Intravitreal Injections in Japanese Patients With Neovascular AMD
Acronym: PINE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1771-101-008
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abicipar pegol (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection
  Interventions: Drug: Abicipar pegol

INTERVENTIONS:
Drug: Abicipar pegol — Abicipar pegol 2 mg administered to the study eye by intravitreal injection
  Other Names: AGN-150998

SUMMARY:
This study will evaluate the safety and to characterize the systemic pharmacokinetics of free and vascular endothelial growth factor (VEGF)-bound abicipar following multiple monthly intravitreal injections of abicipar in Japanese patients with neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female patients
* Presence of active subfoveal and/or juxtafoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD)

Exclusion Criteria:

* History of or active periocular, ocular, or intraocular infection
* Previous use of ocular anti-angiogenic therapy within 1 month (ranibizumab), 6 weeks (pegaptanib), or 2 months (bevacizumab and aflibercept) of Day 1 for the treatment of neovascular AMD or neovascular eye diseases other than AMD
* Macular hemorrhage that involves the center of fovea in the study eye
* Previous use of verteporfin photodynamic therapy (PDT) or previous therapeutic radiation in the region
* Treatment with ocular corticosteroid injections or implants within 6 months in the study eye
* History or evidence of eye surgery: Pars plana vitrectomy, Submacular surgery or other surgical interventions for AMD, Incisional glaucoma surgery or Cataract or refractive surgery within the last 3 months
* AMD or neovascular eye diseases other than AMD in the non-study eye that require anti-VEGF treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Peak Serum Concentration (CMax) for Free and VEGF-Bound Abicipar | Baseline to Week 20
Serum Concentration Immediately before Next Dose (Ctrough) for Free and VEGF-Bound Abicipar | Baseline to Week 20
Time to Cmax (Tmax) for Free and VEGF-Bound Abicipar | Baseline to Week 20
Terminal Elimination Half-Life (t1/2) for Free and VEGF-Bound Abicipar | Baseline to Week 20
Area Under the Serum Concentration-Time Curve from Zero to the End of the Dosing Interval "tau" (AUC0-tau) for Free and VEGF-Bound Abicipar | Baseline to Week 20
Area Under the Serum Concentration-Time Curve from Zero to Infinity (AUC0-inf) for Free and VEGF-Bound Abicipar | Baseline to Week 20

SECONDARY OUTCOMES:
Serum Levels of Anti-abicipar Antibodies | Baseline to Week 20
Percentage of Participants with Treatment Emergent Adverse Events | Baseline to Week 20
Best Corrected Visual Acuity using an Eye Chart | Baseline to Week 20
Percentage of Participants with Change from Baseline in Full Ophthalmic Exam Findings [i.e. Slit Lamp Exam, Intraocular Pressure (IOP) Measurements, Funduscopic Exam] | Baseline to Week 20
Changes from Baseline in General Physical Condition as Measured through General Physical Exam | Baseline to Week 20
Percentage of Participants with Changes from Baseline in Vital Signs (Blood Pressure, Pulse Rate, ECG) | Baseline to Week 20
Percentage of Participants with Change from Baseline in Clinically Relevant Laboratory Values (Serum Chemistry, Hematology, Urinalysis) | Baseline to Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Sutherland, Study Director — Allergan
Locations (5):
- Japan (5):
  - Kimura Eye and Internal Medicine Hospital, Kure, Hiroshima
  - Musashi Dream Clinic, Tennouji-ku, Osaka
  - Takeuchi Eye Clinic, Taito-ku, Tokyo
  - Souseikai Hakata Clinic, Fukuoka
  - Fukushima Medical University Hospital, Fukushima

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com.